CLINICAL TRIAL: NCT07259694
Title: Randomized Controlled Trial on the Effects of Traditional Exercise Programs on the Physical and Mental Health of Hearing-Impaired Individuals
Brief Title: RCT on Traditional Exercise Interventions for Physical and Mental Health in Hearing-Impaired Individuals
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Collaborators: Changchun University (Unknown)
Responsible Party: Principal Investigator, Guang Yang, Prof. Dr., Prof, Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCEE202602
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hearing-Impaired
Keywords: Hearing-Impaired
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Taichi (Experimental)
  Interventions: Behavioral: Taichi
- Baduanjin (Experimental)
  Interventions: Behavioral: Baduanjin
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Taichi — Participants in the Tai Chi group will receive a 12-week simplified 21-form Tai Chi training program. The intervention will consist of supervised sessions conducted three times per week, each lasting approximately 60 minutes. Sessions will include a standardized warm-up, instruction and practice of the 21-form Tai Chi routine, and a brief cool-down period. All training will be delivered by certified Tai Chi instructors experienced in working with individuals with visual impairments. Attendance and adherence will be monitored throughout the intervention period.
  Arms: Taichi
Behavioral: Baduanjin — Participants in the Baduanjin group will undergo a 12-week standardized Baduanjin training program. The intervention will be delivered three times per week, with each supervised session lasting approximately 60 minutes. Training sessions will include a structured warm-up, guided practice of the standardized Baduanjin routine, and a brief cool-down period. All sessions will be led by qualified instructors with experience working with visually impaired individuals. Participant attendance and adherence will be recorded throughout the intervention period.
  Arms: Baduanjin

SUMMARY:
This study aims to investigate the effects and underlying mechanisms of traditional exercise interventions on the physical and mental health of individuals with hearing impairments. A randomized controlled trial will be conducted with 90 participants who will be randomly assigned to one of three groups: a Tai Chi intervention group, a Baduanjin intervention group, or a control group. The Tai Chi group will receive a 12-week simplified 24-form Tai Chi training program, while the Baduanjin group will undergo standardized Baduanjin training. The control group will participate in regular school physical education classes. This study seeks to evaluate the potential health benefits and mechanisms of traditional exercise programs within the hearing-impaired population.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral hearing loss greater than 70 dB.
* No cognitive impairment and able to understand and comply with study procedures.

Exclusion Criteria:

* Neurological disorders affecting balance.
* Severe cardiovascular diseases.
* Significant musculoskeletal or joint disorders.
* Participation in regular exercise training within the past 6 months.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Modified Romberg Test | Month 3
  Assessment of static balance ability using the modified Romberg test administered before and after the intervention.
Y-Balance Test | Month 3
  Evaluation of dynamic balance and lower-limb functional stability using the Y-Balance test at baseline and post-intervention
30-Second Sit-to-Stand Test | Month 3
  Measurement of lower-limb muscular endurance based on the number of sit-to-stand repetitions completed in 30 seconds
Step Test | Month 3
  Assessment of cardiorespiratory fitness using a standardized step test administered at baseline and post-intervention
Reaction Time Test | Month 3
  Evaluation of psychomotor response speed using a computerized reaction time test before and after the intervention
Self-Rated Depression Scale (SDS) | Month 3
  Assessment of depressive symptoms using the SDS at baseline and post-intervention
Self-Rated Anxiety Scale (SAS) | Month 3
  Evaluation of anxiety symptoms using the SAS before and after the intervention
General Self-Efficacy Scale (GSES) | Month 3
  Measurement of perceived self-efficacy using the GSES at baseline and post-intervention.
WHOQOL-BREF | Month 3
  Assessment of quality of life across multiple domains using the WHOQOL-BREF questionnaire administered before and after the intervention
Resting Heart Rate | Month 3
  Measurement of resting heart rate was assessed in a seated position at baseline and post-intervention
Blood Pressure | Month 3
  Assessment of systolic and diastolic blood pressure using a standardized automated device before and after the intervention
Body Mass Index (BMI) | Month 3
  Calculation of BMI based on measured height and weight before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided